CLINICAL TRIAL: NCT06076681
Title: A Phase Ⅰb/Ⅱa, Single-center, Randomized, Open-label Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Preliminary Helicobacter Pylori Eradication Efficacy in Asymptomatic Subjects With Helicobacter Pylori Infection After Multiple Doses of TNP-2198 Capsules Combined With Rabeprazole Sodium Enteric-coated Tablets, or TNP-2198 Capsules Combined With Rabeprazole Sodium Enteric-coated Tablets and Amoxicillin Capsules
Brief Title: A Study to Evaluate Preliminary Helicobacter Pylori Eradication After Multiple Doses of TNP-2198 Capsules Combined With Rabeprazole Sodium Enteric-coated Tablets, or Rabeprazole Sodium Enteric-coated Tablets and Amoxicillin Capsules
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: TenNor Therapeutics (Suzhou) Limited (Industry)
Responsible Party: Sponsor
Organization: TenNor Therapeutics Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TNP-2198-04
Record Dates: First submitted 2023-09-25; First posted 2023-10-11 (Actual); Results first posted 2023-11-22 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Helicobacter Pylori Infection
MeSH Terms: interventions — Rabeprazole; Amoxicillin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group A (Experimental): TNP2198 capsules 200 mg BID + rabeprazole sodium enteric-coated tablets 20 mg BID
  Interventions: Drug: TNP-2198; Drug: Rabeprazole Sodium
- Group B (Experimental): TNP2198 capsules 400 mg BID + rabeprazole sodium enteric-coated tablets 20 mg BID
  Interventions: Drug: TNP-2198; Drug: Rabeprazole Sodium
- Group C (Experimental): TNP2198 capsules 600 mg BID + rabeprazole sodium enteric-coated tablets 20 mg BID
  Interventions: Drug: TNP-2198; Drug: Rabeprazole Sodium
- Group D (Experimental): TNP2198 capsules 400 mg BID + rabeprazole sodium enteric-coated tablets 20 mg BID + amoxicillin capsules 1g BID
  Interventions: Drug: TNP-2198; Drug: Rabeprazole Sodium; Drug: Amoxicillin

INTERVENTIONS:
Drug: TNP-2198 — On Days 1 to 14, all subjects in each group received TNP-2198 capsule within 30 minutes after breakfast and dinner (BID) for 14 consecutive days. On Day 15, the subjects were only administered once within 30 minutes after breakfast.
  Other Names: Rifasutenizol
Drug: Rabeprazole Sodium — On Days 1 to 14, all subjects in each group received rabeprazole within 30 minutes before breakfast and dinner (BID) for 14 consecutive days. On Day 15, the subjects were only administered once within 30 minutes before breakfast.
Drug: Amoxicillin — On Days 1 to 14, all subjects in each group received Amoxicillin capsule within 30 minutes after breakfast and dinner (BID) for 14 consecutive days. On Day 15, the subjects were only administered once within 30 minutes after breakfast.
  Arms: Group D

SUMMARY:
This phase Ⅰb/Ⅱa, single-center, randomized, open-label study was designed to evaluate the safety, tolerability, pharmacokinetics, and preliminary Helicobacter Pylori eradication efficacy in asymptomatic subjects with Helicobacter Pylori infection after multiple doses of TNP-2198 capsules combined with rabeprazole sodium enteric-coated tablets, or TNP-2198 capsules combined with rabeprazole sodium enteric-coated tablets and amoxicillin capsules.

ELIGIBILITY:
Inclusion Criteria:

* Signing the informed consent form and full understanding study contents, process and possible adverse reactions before participation in the study;
* Able to complete the study according to the requirements of the study protocol;
* The subject (including the partner) is willing to take effective contraceptive measures voluntarily without pregnancy plan in the next 6 months;
* Male and female subjects aged 18 to 65 years (inclusive);
* Male subjects' body weight ≥ 50 kg, or female subjects' body weight ≥ 45 kg, with body mass index within the range of 18-30 kg/m2 (inclusive);
* Health condition: no clinically significant history of heart, liver, kidney, digestive tract, nervous system, respiratory system diseases, mental disorders or metabolic abnormalities;
* Normal results or clinically insignificant abnormal results in physical examinations and vital signs;
* Positive result of 14C urea breath test (UBT).
* Clinical laboratory test results are within normal limits or abnormal but without clinical significance as judged by the investigator.

Exclusion Criteria:

* History of Helicobacter Pyloreradication therapy (including participation in other clinical studies of Helicobacter Pylori eradication);
* Average daily consumption of more than 5 cigarettes within 3 months prior to the start of the study;
* History of hypersensitivity to study drug or its excipients, or allergic constitution (allergy to multiple drugs and food);
* History of drug and/or alcohol abuse (mean consumption of ≥ 14 units of alcohol per week: 1 unit = 285 mL of beer, or 25 mL of liquor, or 100 mL of wine);
* Blood donation or massive blood loss (> 450 mL) within 3 months prior to screening;
* Using any drug that changes liver enzyme activity within 28 days prior to screening;
* Taking orally any prescription drug, over-the-counter drug, any vitamin product, or herbal medicine within 14 days prior to screening;
* Taking special diet (including dragon fruit, mango, grapefruit, etc.) or strenuous exercise, or having other factors that affect drug absorption, distribution, metabolism, excretion, etc., within 2 weeks prior to screening;
* Significant changes in diet or exercise habits recently;
* Those who have participated in, or are still participating in clinical studies within 1 months before taking the study drug t;
* With difficulty in swallowing or history of any gastrointestinal diseases that affect drug absorption;
* With any disease that increases the risk of bleeding, such as hemorrhoids, acute gastritis or gastric and duodenal ulcers;
* With clinically significant ECG abnormalities;
* Female subjects who are lactating during the screening period or during the study, or have positive serum pregnancy test results;
* With symptoms or previous history of cardiovascular, digestive, respiratory, urinary, neurological, hematologic, immunological, endocrine system diseases or tumor, or psychiatric diseases;
* Clinically significant abnormalities in clinical laboratory tests, or other clinically significant findings (including but not limited to gastrointestinal, renal, hepatic, neurological, hematological, endocrine, neoplastic, pulmonary, immunological, psychiatric, or cardiovascular disease);
* Those who have positive tests results of viral hepatitis (including hepatitis B and C), HIV antibody, treponema pallidum antibody (additional RPR test is required for those with positive treponema pallidum antibody);
* Acute illness occurs or concomitant medication is used from the date of signing the informed consent to the date prior to study medication;
* Consumption of chocolate, any caffeine- or xanthine-containing food or drink within 48 hours prior to taking the study drug;
* Consumption of any alcoholic product within 48 hours prior to taking the study drug;
* Those who have positive test result of urine drug screening or history of drug abuse or drug addiction within the past 5 years;
* Those who have other conditions that, in the opinion of the investigator, make participation in this study inappropriate.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-09-27 (Actual); Primary Completion 2022-01-06 (Actual); Study Completion 2022-01-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: TenNor Clinical Trials, Study Director — TenNor
Locations (1):
- The First Hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li X, Liu Y, Wang M, Gao L, Liu J, Zhang H, Wu M, Chen H, Lou J, Wang J, Chen J, Geng G, Ma Z, Ding Y. Safety, pharmacokinetics, and efficacy of rifasutenizol, a novel dual-targeted antibacterial agent in healthy participants and patients in China with Helicobacter pylori infection: four randomised clinical trials. Lancet Infect Dis. 2024 Jun;24(6):650-664. doi: 10.1016/S1473-3099(24)00003-3. Epub 2024 Feb 12. PMID 38359854

RESULTS

PARTICIPANT FLOW:
Groups:
- Group A: TNP-2198 capsules 200 mg BID + rabeprazole sodium enteric-coated tablets 20 mg BID
  On Days 1 to 14, all subjects received TNP-2198 capsules(200mg) and rabeprazole sodium enteric-coated tablets (20 mg) within 30 minutes after breakfast and dinner (BID) for 14 consecutive days. On Day 15, the subjects were only administered once within 30 minutes after breakfast.
- Group B: TNP-2198 capsules 400 mg BID + rabeprazole sodium enteric-coated tablets 20 mg BID
  On Days 1 to 14, all subjects received TNP-2198 capsules(400mg) and rabeprazole sodium enteric-coated tablets (20 mg) within 30 minutes after breakfast and dinner (BID) for 14 consecutive days. On Day 15, the subjects were only administered once within 30 minutes after breakfast.
- Group C: TNP-2198 capsules 600 mg BID + rabeprazole sodium enteric-coated tablets 20 mg BID
  On Days 1 to 14, all subjects received TNP-2198 capsules(600 mg) and rabeprazole sodium enteric-coated tablets (20 mg) within 30 minutes after breakfast and dinner (BID) for 14 consecutive days. On Day 15, the subjects were only administered once within 30 minutes after breakfast.
- Group D: TNP-2198 capsules 400 mg BID + rabeprazole sodium enteric-coated tablets 20 mg BID + amoxicillin capsules 1g BID
  On Days 1 to 14, all subjects received TNP-2198 capsules(400mg), rabeprazole sodium enteric-coated tablets(20mg) and Amoxicillin capsules(1g) within 30 minutes after breakfast and dinner (BID) for 14 consecutive days. On Day 15, the subjects were only administered once within 30 minutes after breakfast.
Period: Overall Study
Arm/Group | Group A | Group B | Group C | Group D
Started | 10 | 10 | 10 | 10
Completed | 10 | 10 | 10 | 10
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Group C | Group D | Total
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 10 | 10 | 40
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.8 (9.09) | 38.3 (10.31) | 41.4 (6.36) | 40.6 (10.73) | 40.0 (8.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 3 | 6 | 20
  Male | 5 | 4 | 7 | 4 | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 10 | 10 | 10 | 10 | 40
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: The Eradication Rate of Helicobacter Pylori Infection
Description: Eradication rate of H. pylori is defined as negative urea breath test result.
Time Frame: Urea breath test is assessed 4-6 weeks after the treatment (Day 44~ Day 50)
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B | Group C | Group D
Number analyzed (Participants) | 10 | 10 | 10 | 10
Participants | 0 | 3 | 4 | 8

ADVERSE EVENTS:
Time Frame: Day 1 to Day 17
Arm/Group | Group A | Group B | Group C | Group D
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 6/10 | 8/10 | 5/10 | 8/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A (N=10) | Group B (N=10) | Group C (N=10) | Group D (N=10)
Blood Creatinine Increased (Investigations) | 3 (4) | 1 (1) | 1 (2) | 1 (2)
Alanine aminotransferase(AST)increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (3) | 2 (2) | 1 (1) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0) | 2 (2)
White blood cell count decreased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Neutrophil count decreased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-20): https://cdn.clinicaltrials.gov/large-docs/81/NCT06076681/Prot_SAP_000.pdf